CLINICAL TRIAL: NCT01023308
Title: A Multicenter, Randomized, Double Blind, Placebo Controlled Phase III Study of Panobinostat in Combination With Bortezomib and Dexamethasone in Patients With Relapsed Multiple Myeloma
Brief Title: Panobinostat or Placebo With Bortezomib and Dexamethasone in Patients With Relapsed Multiple Myeloma
Acronym: PANORAMA-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLBH589D2308; 2009-015507-52 (EudraCT Number)
Record Dates: First submitted 2009-11-30; First posted 2009-12-02 (Estimated); Results first posted 2015-10-23 (Estimated); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Multiple Myeloma
Keywords: Myeloma; DACi; Bortezomib; Combination; Panobinostat; LBH589D; relapsed; Velcade®; Combination,
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell; Recurrence | interventions — Panobinostat; Bortezomib; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Panobinostat + Bortezomib + Dexamethasone (Experimental)
  Interventions: Drug: Panobinostat; Drug: Bortezomib; Drug: Dexamethasone
- Placebo + Bortezomib + Dexamethasone (Placebo Comparator)
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Placebo

INTERVENTIONS:
Drug: Panobinostat — Panobinostat was administered 3x week ( 2 weeks on 1 week off)
  Other Names: LBH589
  Arms: Panobinostat + Bortezomib + Dexamethasone
Drug: Bortezomib — Bortezomib was administered 2 x week ( 2weeks on 1 week off)
  Other Names: (Velcade®)
Drug: Dexamethasone — Dexamethasone was adminstered on day of Bortezomib and the day after Bortezomib administration
Drug: Placebo — Placebo was administered 3x week ( 2 weeks on 1 week off)
  Arms: Placebo + Bortezomib + Dexamethasone

SUMMARY:
Panobinostat (LBH589) is a highly potent pan-deacetylase inhibitor (pan-DACi), inclusive of HDAC6, which disrupts aggresome function, promotes accumulation of cytotoxic misfolded protein aggregates and triggers myeloma cell death. Combination of pan-DAC and protease inhibition by co-treatment with panobinostat (PAN) and bortezomib (BTZ) has demonstrated synergistic cytotoxicity in vitro and in vivo in pre-clinical experiments. Furthermore, clinical experience in advanced multiple myeloma (MM) patients treated by oral panobinostat and i.v bortezomib ± dexamethasone showed very encouraging results for efficacy and manageable toxicity profile.

Given the medical need for improved treatment strategies for patients with previously treated and relapsed MM, the purpose of this prospective, multinational, randomized, double-blind, placebo-controlled, parallel group Phase III study is to compare the results in progression-free survival of 2 combination therapies, panobinostat with bortezomib and dexamethasone or placebo with bortezomib and dexamethasone, in patients with previously treated MM whose disease has recurred or progressed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a previous diagnosis of multiple myeloma.
2. Patient requires retreatment for multiple myeloma
3. Patient has measurable M component in serum or urine at study screening

Exclusion Criteria:

1. Patient who has progressed under all prior lines of anti MM therapy
2. Patient who has been treated by bortezomib before, and did not reach at least a minor response under this therapy, or progressed under it or within 60 days of last dose
3. Patient has shown intolerance to bortezomib or to dexamethasone or components of these drugs or has any contraindication to one or the other drug , following locally applicable prescribing information
4. Patient received prior treatment with DAC inhibitors including panobinostat
5. Patient has impaired cardiac function, or a prolonged QTc interval at screening ECG
6. Patient taking medications with relative risk of prolonging the QT interval or inducing Torsade de pointes
7. Female patient who is pregnant or breast feeding or with childbearing potential and not willing to use a double method of contraception up to 3 months after the end of study treatment. Male patient who is not willing to use a barrier method of contraception up to 3 months after the end of study treatment.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 767 (Actual)
Dates: Start 2009-12-21 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2015-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (192):
- United States (37):
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Concord, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, San Diego, California
  - Novartis Investigative Site, Stanford, California
  - Novartis Investigative Site, Boca Raton, Florida
  - Novartis Investigative Site, Lake Worth, Florida
  - Novartis Investigative Site, Miami Shores, Florida
  - Novartis Investigative Site, Athens, Georgia
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Marywood, Illinois
  - Novartis Investigative Site, Quincy, Illinois
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Rockville, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Southfield, Michigan
  - Novartis Investigative Site, Edina, Minnesota
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Columbia, Missouri
  - Novartis Investigative Site, East Orange, New Jersey
  - Novartis Investigative Site, Mount Kisco, New York
  - Novartis Investigative Site, Durham, North Carolina
  - Novartis Investigative Site, Bismarck, North Dakota
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Middletown, Ohio
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, East Providence, Rhode Island
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Amarillo, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Kennewick, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Walla Walla, Washington
  - Novartis Investigative Site, Morgantown, West Virginia
- Argentina (3):
  - Novartis Investigative Site, La Plata, Buenos Aires
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Córdoba
- Australia (6):
  - Novartis Investigative Site, St Leonards, New South Wales
  - Novartis Investigative Site, Herston, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Franston, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
  - Novartis Investigative Site, Perth, Western Australia
- Austria (2):
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Vienna
- Belgium (3):
  - Novartis Investigative Site, Jette, Brussels Capital
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Hasselt
- Brazil (5):
  - Novartis Investigative Site, Brasília, Federal District
  - Novartis Investigative Site, Rio de Janeiro, Rio de Janeiro
  - Novartis Investigative Site, Barretos, São Paulo
  - Novartis Investigative Site, Campinas, São Paulo
  - Novartis Investigative Site, São Paulo, São Paulo
- Canada (5):
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Greenfield Park, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- China (9):
  - Novartis Investigative Site, Beijing, Beijing Municipality
  - Novartis Investigative Site, Nanning, Guangxi
  - Novartis Investigative Site, Nanjing, Jiangsu
  - Novartis Investigative Site, Suzhou, Jiangsu
  - Novartis Investigative Site, Chengdu, Sichuan
  - Novartis Investigative Site, Tianjin, Tianjin Municipality
  - Novartis Investigative Site, Hangzhou, Zhejiang
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Shanghai
- Czechia (3):
  - Novartis Investigative Site, Brno-Bohunice, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Olomouc, CZE
- Denmark (5):
  - Novartis Investigative Site, Aalborg
  - Novartis Investigative Site, Aarhus
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Odense
  - Novartis Investigative Site, Vejle
- Egypt (2):
  - Novartis Investigative Site, Alexandria
  - Novartis Investigative Site, Giza
- Finland (2):
  - Novartis Investigative Site, HUS Helsinki
  - Novartis Investigative Site, Turku
- France (9):
  - Novartis Investigative Site, Blois
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Limoges
  - Novartis Investigative Site, Nantes
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Vandœuvre-lès-Nancy
- Germany (17):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Bamberg
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bremen
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Duisburg
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Jena
  - Novartis Investigative Site, Kiel
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Rostock
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg
- Greece (2):
  - Novartis Investigative Site, Thessaloniki, GR
  - Novartis Investigative Site, Athens
- Hong Kong (3):
  - Novartis Investigative Site, New Territories, Hong Kong
  - Novartis Investigative Site, Hong Kong
  - Novartis Investigative Site, Hong Kong SAR
- Israel (4):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Kfar Saba
  - Novartis Investigative Site, Petah Tikva
  - Novartis Investigative Site, Ramat Gan
- Italy (11):
  - Novartis Investigative Site, San Giovanni Rotondo, FG
  - Novartis Investigative Site, Lecce, LE
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Pescara, PE
  - Novartis Investigative Site, Pisa, PI
  - Novartis Investigative Site, Pavia, PV
  - Novartis Investigative Site, Reggio Calabria, RC
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Pagani, SA
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Napoli
- Japan (13):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Ōgaki, Gifu
  - Novartis Investigative Site, Shibukawa, Gunma
  - Novartis Investigative Site, Kure, Hiroshima
  - Novartis Investigative Site, Higashiibaraki-gun, Ibaraki
  - Novartis Investigative Site, Okayama, Okayama-ken
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Shibuya City, Tokyo
  - Novartis Investigative Site, Hiroshima
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Osaka
- Novartis Investigative Site, Beirut, Lebanon
- Novartis Investigative Site, San Luis Potosí City, Mexico
- Netherlands (2):
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Utrecht
- Norway (6):
  - Novartis Investigative Site, Bergen
  - Novartis Investigative Site, Fredrikstad
  - Novartis Investigative Site, Kristiansand
  - Novartis Investigative Site, Oslo
  - Novartis Investigative Site, Skien
  - Novartis Investigative Site, Trondheim
- Novartis Investigative Site, Warsaw, Poland
- Russia (2):
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Saratov
- Novartis Investigative Site, Singapore, Singapore
- South Africa (2):
  - Novartis Investigative Site, Parktown
  - Novartis Investigative Site, Pretoria
- South Korea (7):
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Jeollanam-do, Jeollanam-do
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul
  - Novartis Investigative Site, Taegu
- Spain (10):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Donostia / San Sebastian, Basque Country
  - Novartis Investigative Site, Salamanca, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Pamplona, Navarre
  - Novartis Investigative Site, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
- Sweden (5):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Linköping
  - Novartis Investigative Site, Luleå
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Taiwan (4):
  - Novartis Investigative Site, Kaohsiung City
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- Novartis Investigative Site, Bangkok, Thailand
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
- United Kingdom (5):
  - Novartis Investigative Site, Aberdeen, Scotland
  - Novartis Investigative Site, Glasgow, Scotland
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Wolverhampton

REFERENCES:
- [Derived] San-Miguel JF, Hungria VT, Yoon SS, Beksac M, Dimopoulos MA, Elghandour A, Jedrzejczak WW, Gunther A, Nakorn TN, Siritanaratkul N, Schlossman RL, Hou J, Moreau P, Lonial S, Lee JH, Einsele H, Sopala M, Bengoudifa BR, Binlich F, Richardson PG. Overall survival of patients with relapsed multiple myeloma treated with panobinostat or placebo plus bortezomib and dexamethasone (the PANORAMA 1 trial): a randomised, placebo-controlled, phase 3 trial. Lancet Haematol. 2016 Nov;3(11):e506-e515. doi: 10.1016/S2352-3026(16)30147-8. Epub 2016 Oct 14. PMID 27751707
- [Derived] San-Miguel JF, Einsele H, Moreau P. The Role of Panobinostat Plus Bortezomib and Dexamethasone in Treating Relapsed or Relapsed and Refractory Multiple Myeloma: A European Perspective. Adv Ther. 2016 Nov;33(11):1896-1920. doi: 10.1007/s12325-016-0413-7. Epub 2016 Sep 27. PMID 27677481
- [Derived] Richardson PG, Hungria VT, Yoon SS, Beksac M, Dimopoulos MA, Elghandour A, Jedrzejczak WW, Guenther A, Nakorn TN, Siritanaratkul N, Schlossman RL, Hou J, Moreau P, Lonial S, Lee JH, Einsele H, Sopala M, Bengoudifa BR, Corrado C, Binlich F, San-Miguel JF. Panobinostat plus bortezomib and dexamethasone in previously treated multiple myeloma: outcomes by prior treatment. Blood. 2016 Feb 11;127(6):713-21. doi: 10.1182/blood-2015-09-665018. Epub 2015 Dec 2. PMID 26631116
- [Derived] San-Miguel JF, Hungria VT, Yoon SS, Beksac M, Dimopoulos MA, Elghandour A, Jedrzejczak WW, Gunther A, Nakorn TN, Siritanaratkul N, Corradini P, Chuncharunee S, Lee JJ, Schlossman RL, Shelekhova T, Yong K, Tan D, Numbenjapon T, Cavenagh JD, Hou J, LeBlanc R, Nahi H, Qiu L, Salwender H, Pulini S, Moreau P, Warzocha K, White D, Blade J, Chen W, de la Rubia J, Gimsing P, Lonial S, Kaufman JL, Ocio EM, Veskovski L, Sohn SK, Wang MC, Lee JH, Einsele H, Sopala M, Corrado C, Bengoudifa BR, Binlich F, Richardson PG. Panobinostat plus bortezomib and dexamethasone versus placebo plus bortezomib and dexamethasone in patients with relapsed or relapsed and refractory multiple myeloma: a multicentre, randomised, double-blind phase 3 trial. Lancet Oncol. 2014 Oct;15(11):1195-206. doi: 10.1016/S1470-2045(14)70440-1. Epub 2014 Sep 18. PMID 25242045
- See also: Related Info — http://NovartisClinicalTrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Panobinostat + Bortezomib: Panobinostat was given 20 mg hard gelatin capsules . Bortezomib was given at 1.3 mg/m2 as a 3 to 5 second bolus intravenous (IV)injection. Dexamethasone was given as an oral dose of 20 mg/day.
- Placebo + Bortezomib: Placebo was given as a hard gelatin capsule in the image of Panobinostat . Bortezomib was given at 1.3 mg/m2 as a 3 to 5 second bolus intravenous (IV) injection. Dexamethasone was given as an oral dose of 20 mg/day.
Period: Overall Study
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Started | 387 | 381
Completed | 102 (completed all planned cycles of study treatment as per protocol) | 102 (completed all planned cycles of study treatment as per protocol)
Not Completed | 285 | 279
Not completed — Abnormal test proceedure results | 3 | 8
Not completed — Administrative problems | 2 | 1
Not completed — Adverse Event | 130 | 66
Not completed — Death | 21 | 17
Not completed — Disease progression | 82 | 153
Not completed — New Cancer therapy | 4 | 7
Not completed — Protocol Violation | 3 | 4
Not completed — Untreated | 5 | 5
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 34 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib | Total
Number analyzed (Participants) | 387 | 381 | 768
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.4 (9.34) | 61.8 (9.43) | 62.1 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 185 | 176 | 361
  Male | 202 | 205 | 407
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 249 | 250 | 499
  Asian | 128 | 104 | 232
  Black | 5 | 17 | 22
  Other | 5 | 10 | 15

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival Events in Patients Treated With Panobinostat in Combination With Bortezomib and Dexamethasone vs. Patients Treated by Placebo in Combination With Bortezomib and Dexamethasone.
Time Frame: 45 months
Measure: Number; unit: number of events
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 387 | 381
number of events | 207 | 260

2. Primary Outcome: Progression Free Survival in Patients Treated With Panobinostat in Combination With Bortezomib and Dexamethasone vs. Patients Treated by Placebo in Combination With Bortezomib and Dexamethasone.
Time Frame: 45 months
Population: Full Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 387 | 381
months | 11.99 [10.32 to 12.94] | 8.80 [7.56 to 9.23]

3. Secondary Outcome: Overall Survival in Patients Treated With Panobinostat in Combination With Bortezomib and Dexamethasone vs. Patients Treated by Placebo in Combination With Bortezomib and Dexamethasone
Description: Number of OS events
Time Frame: 45 months
Measure: Number; unit: Number of OS events
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 387 | 381
Number of OS events | 134 | 152

4. Secondary Outcome: Overall Survival in Patients Treated With Panobinostat in Combination With Bortezomib and Dexamethasone vs. Patients Treated by Placebo in Combination With Bortezomib and Dexamethasone
Description: survival time in months
Time Frame: 45 months
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 387 | 381
months | 40.28 [35.02 to 44.81] | 35.78 [28.98 to 40.64]

5. Secondary Outcome: Overall Response Rate in Patients Treated With Panobinostat in Combination With Bortezomib and Dexamethasone vs. Patients Treated by Placebo in Combination With Bortezomib and Dexamethasone.
Description: Best overall response based on mEBMT criteria per investigator assessment
Time Frame: 45 months
Measure: Number; unit: % participants with response
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 387 | 381
% participants with response | 60.7 | 54.6

6. Secondary Outcome: Time to Response Per Investigator Assessment (mEBMT Criteria) of Response Patients Treated With Panobinostat in Combination With Bortezomib and Dexamethasone vs. Patients Treated by Placebo in Combination With Bortezomib and Dexamethasone.
Time Frame: 45 months
Measure: Median (95% Confidence Interval); unit: time to response in months
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 387 | 381
time to response in months | 1.51 [1.41 to 1.64] | 2.00 [1.61 to 2.79]

7. Secondary Outcome: Duration of Response Per Investigator Assessment (mEBMT Criteria) Patients Treated With Panobinostat in Combination With Bortezomib and Dexamethasone vs. Patients Treated by Placebo in Combination With Bortezomib and Dexamethasone.
Time Frame: 45 months
Measure: Median (95% Confidence Interval); unit: duration of response in months
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 387 | 381
duration of response in months | 13.14 [11.76 to 14.92] | 10.87 [9.23 to 11.76]

8. Secondary Outcome: Time to Progression/Relapse Per Investigator Assessment (mEBMT Criteria) Patients Treated With Panobinostat in Combination With Bortezomib and Dexamethasone vs. Patients Treated by Placebo in Combination With Bortezomib and Dexamethasone.
Time Frame: 45 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 387 | 381
months | 12.71 [11.30 to 14.06] | 8.54 [7.66 to 9.72]

9. Secondary Outcome: European Organization for Research and Treatment of Cancer Multiple Myeloma Module (EORTC) QLQ-MY20-Change From Baseline by Treatment Group
Description: Higher values in the disease symptoms and side effects of treatment scores indicate worsening. Higher scores in the future perspective and body image scores indicate improvement. LS Means and SEM are estimated from the repeated measures model. Following factors and covariates are included in the repeated measurement model: time, treatment, treatment by time interaction, number of prior lines of anti-MM therapy (1/ 2 and 3), prior use of BTZ (Yes/ No), baseline score.Disease Symptom is the sum of 20 questions, total score ranges from 0 (best possible outcome) to 100 (worst possible outcome)", All subscales of EORTC QLQ-MY20 have the same score range of 0 -100. Decrease in symptom scores from baseline indicate improvement in symptoms.
Time Frame: 12, 24 and 48 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 387 | 381
score on a scale
  Disease Symptom wk 12 change baseline (n=215,243) | -4.795 [-6.76 to -2.83] | -4.865 [-6.75 to -2.98]
  Disease Symptom wk 24 change baseline (n=148,177) | -4.401 [-6.53 to -2.27] | -6.797 [-8.79 to -4.81]
  Disease Symptom wk 48 change baseline (n=37,26) | -2.836 [-6.76 to -1.084] | -6.626 [-11.1 to -2.12]
  Side effects of treatment wk 12 chge (n=213,242) | 8.162 [6.510 to 9.814] | 5.524 [3.933 to 7.115]
  Side effects of treatment wk 24 chge (n=148,175) | 9.016 [6.955 to 11.08] | 7.731 [5.795 to 9.668]
  Side effects of treatment wk 48 chge (n=37,26) | 3.357 [0.442 to 6.273] | 3.654 [0.352 to 6.956]
  Future perspective wk 12 chge (n=214,242) | 5.319 [2.893 to 7.744] | 6.194 [3.854 to 8.533]
  Future perspective wk 24 chge (n=148,176) | 3.877 [0.977 to 6.778] | 5.839 [3.103 to 8.575]
  Future perspective wk 48 chge (n=37,26) | 4.331 [-.142 to 8.804] | 6.951 [1.807 to 12.10]
  Body image wk 12 chge (n=213,240) | -7.178 [-10.5 to -3.87] | -6.22 [-9.41 to -3.03]
  Body image wk 24 chge (n=147,175) | -11.463 [-15.3 to -7.66] | -7.358 [-10.9 to -3.81]
  Body image wk 48 chge (n=37,26) | -2.161 [-7.73 to 3.410] | -4.666 [-11.1 to 1.729]

10. Secondary Outcome: European Organization for Research and Treatment of Cancer Multiple Myeloma Module (EORTC ) QLQ-C30 - Summary Statistics by Treatment Group
Description: The EORTC QLQ-C30 measures functional dimensions (physical, role, emotional, cognitive, and social), three multi-item symptom scales (fatigue, nausea/vomiting, and pain), six single-item symptom scales (dyspnea, sleep disturbance, appetite loss, constipation, diarrhea and financial impact) and a global health status/QoL scale. Disease Symptom is the sum of 30 questions, total score ranges from 0 (best possible outcome) to 100 (worst possible outcome)", All subscales of EORTC QLQ-C30 have the same score range of 0 -100. For global health status and other functional scales,an increase from baseline indicates improvement of QoL. Whereas for symptoms scales, fatigue, dyspnea, insomnia, appetite loss, constipation and diarrhea, decrease in scores from baseline indicate improvement in symptoms.
Time Frame: 12, 24 and 48 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 387 | 381
score on a scale
  Global health wk 12 change baseline (n=216,239) | -9.853 [-12.50 to -7.20] | -4.044 [-6.60 to -1.49]
  Global health wk 24 change baseline (n=150,176) | -7.867 [-10.7 to -5.08] | -1.518 [-4.11 to -1.075]
  Global health wk 48 change baseline (n=38,26) | -2.986 [-7.21 to 1.237] | 4.345 [-0.416 to 9.106]
  Physical functioning wk 12 chge (n=217,242) | -9.67 [-12.00 to -7.38] | -5.393 [-76.3 to -3.16]
  Physical functioning wk 24 chge (n=151,177) | -9.516 [-12.20 to -7.38] | -6.456 [-8.98 to -3.93]
  Physical functioning wk 48 chge (n=38,26) | -2.88 [-6.41 to 0.651] | 2.037 [-2.07 to 6.147]
  Role functioning wk 12 chge (n=215,237) | -11.159 [-14.6 to -7.74] | -6.762 [-10.1 to -3.45]
  Role functioning wk 24 chge (n=150,176) | -11.875 [-15.7 to -8.01] | -11.263 [-14.9 to -7.61]
  Role functioning wk 48 chge (n=38,26) | -5.927 [-11.4 to -0.424] | -0.401 [-6.73 to 5.924]
  Cognitive functioning wk 12 chge (n=216,240) | -4.464 [-6.89 to -2.04] | -1.023 [-3.36 to 1.318]
  Cognitive functioning wk 24 chge (n=149,176) | -6.053 [-8.87 to -3.24] | -3.542 [-6.22 to -0.865]
  Cognitive functioning wk 48 chge (n=38,26) | -5.568 [-9.79 to -1.34] | -4.042 [-8.99 to 0.902]
  Social functioning wk 12 chge (n=216,240) | -8.502 [-11.6 to -5.44] | -3.991 [-6.97 to 1.02]
  Social functioning wk 24 chge (n=148,171) | -8.925 [-12.4 to -5.42] | -6.338 [-9.66 to -3.02]
  Social functioning wk 48 chge (n=37,26) | -6.104 [-11.0 to -1.22] | 4.617 [-0.930 to 10.16]
  Fatigue wk 12 chge (n=217,241) | 15.122 [12.27 to 17.98] | 7.939 [5.174 to 10.70]
  Fatigue wk 24 chge (n=151,176) | 12.677 [9.419 to 15.94] | 9.203 [6.136 to 12.27]
  Fatigue wk 48 chge(n=38,26) | 4.646 [0.086 to 9.206] | -2.625 [-7.88 to 2.628]
  Dyspnea wk 12 chge (n=217,240) | 13.964 [10.60 to 17.33] | 6.266 [3.012 to 9.521]
  Dyspnea wk 24 chge (n=151,177) | 7.939 [4.639 to 11.24] | 5.308 [2.221 to 8.394]
  Dyspnea wk 48 chge (n=38,26) | 4.118 [-1.58 to 9.813] | 2.82 [-3.88 to 9.523]
  Insomnia wk 12 chge (n=216,239) | 6.283 [2.851 to 9.715] | 7.625 [4.331 to 10.92]
  Insomnia wk 24 chge (n=149,176) | 10.023 [6.038 to 14.01] | 6.104 [2.381 to 9.827]
  Insomnia wk 48 chge (n=38,26) | -2.464 [-8.74 to 3.811] | -3.442 [-10.9 to 4.017]
  Appetite loss wk 12 chge (n=217,239) | 15.167 [11.60 to 18.74] | 5.383 [1.925 to 8.841]
  Appetite loss wk 24 chge (n=151,176) | 16.574 [12.39 to 20.76] | 5.861 [1.918 to 9.804]
  Appetite loss wk 48 chge (n=38,26) | 3.999 [-2.08 to 10.07] | -2.963 [-9.99 to 4.061]
  Constipation wk 12 chge (n=215,240) | 4.135 [0.667 to 7.603] | 6.42 [3.104 to 9.735]
  Constipation wk 24 chge (n=151,177) | -0.153 [-3.64 to 3.337] | 0.524 [-2.73 to 5.782]
  Constipation wk 48 chge (n=38,25) | -0.358 [-5.57 to 4.851] | -0.946 [-7.26 to 5.373]
  Diarrhea wk 12 chge (n=217,241) | 18.888 [15.04 to 22.74] | 10.206 [6.452 to 13.96]
  Diarrhea wk 24 chge (n=150,177) | 23.163 [18.46 to 27.87] | 16.406 [11.98 to 20.83]
  Diarrhea wk 48 chge (n=38,26) | 20.48 [14.02 to 26.94] | 10.996 [3.422 to 18.57]

11. Secondary Outcome: Functional Assessment of Chronic Illness Therapy (FACIT) Measurement System : FACT/GOG-NTX-Change From Baseline by Treatment Group
Description: Chronic Illness Therapy (FACIT) Measurement System and focuses on four general quality of life domains for physical well being, functional well-being, social/family well-being, and emotional well-being, and includes additional items to characterize treatment-related neurotoxicity. Higher subscales/total scores represent higher QOL. In the case of the neurotoxicity subscale, lower scores correspond to higher neurotoxicity. The recall period referenced in the questionnaire is the past 7 days.Ranges for FACT-G subscales are as follows:.PWB, scale 0 -28, , NtxS scale 0-44, FACT/GOG-Ntx trial outcome index scale is 0-100 and FACT-G scale is also scaled 0-100. An increase from baseline in these scores indicate improvement.
Time Frame: 12, 24 and 48 weeks
Population: Full Analysis Set
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Panobinostat + Bortezomib | Placebo + Bortezomib
Number analyzed (Participants) | 387 | 381
score on a scale
  Neurotoxicity wk 12 change baseline (n=212,240) | -4.481 [-5.33 to -3.63] | -3.337 [-4.17 to -2.50]
  Neurotoxicity wk 24 change baseline (n=148,174) | -4.564 [-5.49 to -3.64] | -4.739 [-5.61 to -3.86]
  Neurotoxicity wk 48 change baseline (n=35,26) | -3.158 [-4.52 to -1.79] | -2.133 [-3.64 to -0.627]
  Physical wellbeing wk 12 chge (n=215,240) | -3.29 [-3.94 to -2.64] | -1.952 [-2.58 to -1.32]
  Physical wellbeingwk 24 chge (n=150,176) | -3.044 [-3.74 to -2.35] | -2.259 [-2.92 to -1.60]
  Physical wellbeing wk 48 chge (n=38,26) | -2.037 [-3.08 to -0.992] | 0.203 [-1.03 to 1.439]
  Trial Outcomes wk 12 chge (n=209,236) | -10.573 [-12.2 to -8.86] | -6.874 [-8.55 to -5.19]
  Trial Outcomes wk 24 chge (n=148,173) | -9.84 [-11.7 to -7.98] | -8.894 [-10.7 to -7.13]
  Trial Outcomes wk 48 chge (n=35,26) | -6.633 [-9.28 to -3.98] | -2.821 [-5.76 to 0.122]
  FACT-G Total wk 12 chge (n=213,240) | -6.658 [-8.23 to -5.09] | -4.106 [-5.64 to -2.57]
  FACT-G Totalwk 24 chge (n=147,175) | -6.076 [-7.84 to -4.31] | -4.609 [-6.30 to -2.92]
  FACT-G Total wk 48 chge (n=37,26) | -2.704 [-5.29 to -0.118] | -1.435 [-4.42 to 1.547]
  FACT/GOGNTX Total wk 12 chge (n=206,230) | -11.176 [-13.3 to -9.03] | -7.524 [-9.64 to -5.41]
  FACT/GOGNTX Total wk 24 chge (n=146,172) | -10.581 [-12.9 to -8.23] | -9.179 [-9.64 to -5.41]
  FACT/GOGNTX Total wk 48 chge (n=35,26) | -5.871 [-9.24 to -2.50] | -3.151 [-6.92 to 0.614]

ADVERSE EVENTS:
Time Frame: Safety Set consists of all patients who received at least one dose of any component of the study treatment. 10 patients were randomized but did not receive treatment. 6 patients from PAN+BTZ+Dex and 4 patients from PBO+BTZ+Dex
Groups:
- PAN+BTZ: Panobinostat was given 20 mg hard gelatin capsules . Bortezomib was given at 1.3 mg/m2 as a 3 to 5 second bolus intravenous (IV)injection. Dexamethasone was given as an oral dose of 20 mg/day.
- PBO+BTZ: Placebo was given as a hard gelatin capsule in the image of Panobinostat . Bortezomib was given at 1.3 mg/m2 as a 3 to 5 second bolus intravenous (IV) injection. Dexamethasone was given as an oral dose of 20 mg/day..
Arm/Group | PAN+BTZ | PBO+BTZ
Serious Adverse Events (participants affected / at risk) | 228/381 | 157/377
Other Adverse Events (participants affected / at risk) | 379/381 | 366/377
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PAN+BTZ (N=381) | PBO+BTZ (N=377)
Anaemia (Blood and lymphatic system disorders) | 14 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 1
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Monocytosis (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 28 | 8
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 2 | 2
Atrial fibrillation (Cardiac disorders) | 4 | 2
Atrial flutter (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 2 | 2
Cardiac failure (Cardiac disorders) | 1 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 2 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Conjunctivitis (Eye disorders) | 1 | 0
Exophthalmos (Eye disorders) | 1 | 0
Optic ischaemic neuropathy (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 3 | 0
Constipation (Gastrointestinal disorders) | 3 | 3
Diarrhoea (Gastrointestinal disorders) | 43 | 9
Dysphagia (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 0
Gastritis (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 2 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 5 | 3
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 2 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 7 | 0
Necrotising oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 2 | 1
Peritoneal necrosis (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 12 | 3
Asthenia (General disorders) | 15 | 6
Chest discomfort (General disorders) | 1 | 1
Chills (General disorders) | 1 | 0
Fatigue (General disorders) | 11 | 2
General physical health deterioration (General disorders) | 2 | 0
Generalised oedema (General disorders) | 1 | 0
Hypothermia (General disorders) | 0 | 2
Multi-organ failure (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 3
Oedema peripheral (General disorders) | 1 | 0
Pyrexia (General disorders) | 16 | 11
Spinal pain (General disorders) | 0 | 1
Sudden death (General disorders) | 1 | 1
Biliary dyskinesia (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatomegaly (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Acute tonsillitis (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Aspergillosis (Infections and infestations) | 1 | 0
Atypical pneumonia (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bacteriuria (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 3 | 2
Bronchopneumonia (Infections and infestations) | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 1
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Cytomegalovirus colitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Device related sepsis (Infections and infestations) | 1 | 0
Disseminated tuberculosis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Enteritis infectious (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 7 | 2
Gastroenteritis salmonella (Infections and infestations) | 2 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Haemophilus sepsis (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 3 | 1
Herpes zoster (Infections and infestations) | 4 | 5
Infection (Infections and infestations) | 5 | 2
Influenza (Infections and infestations) | 1 | 1
Lobar pneumonia (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 3
Lung infection (Infections and infestations) | 2 | 2
Nasopharyngitis (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 2
Neutropenic sepsis (Infections and infestations) | 2 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 1 | 0
Periodontitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 1
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 56 | 40
Pneumonia bacterial (Infections and infestations) | 0 | 2
Pneumonia fungal (Infections and infestations) | 2 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Pneumonia influenzal (Infections and infestations) | 2 | 1
Pneumonia pneumococcal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 1
Respiratory tract infection (Infections and infestations) | 4 | 2
Salmonellosis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 9 | 7
Septic shock (Infections and infestations) | 9 | 2
Sinusitis (Infections and infestations) | 1 | 1
Skin infection (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Urinary tract infection (Infections and infestations) | 8 | 4
Varicella (Infections and infestations) | 1 | 0
Viral haemorrhagic cystitis (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 3 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood creatinine increased (Investigations) | 1 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
Blood potassium decreased (Investigations) | 0 | 1
Blood pressure decreased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 2 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 2
General physical condition abnormal (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 4 | 0
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 4 | 2
Dehydration (Metabolism and nutrition disorders) | 11 | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypochloraemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Hypophagia (Metabolism and nutrition disorders) | 2 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Altered state of consciousness (Nervous system disorders) | 1 | 0
Autonomic neuropathy (Nervous system disorders) | 1 | 0
Brain compression (Nervous system disorders) | 0 | 1
Brain injury (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Central nervous system haemorrhage (Nervous system disorders) | 0 | 1
Central nervous system necrosis (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 2
Cerebrovascular accident (Nervous system disorders) | 3 | 0
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Cranial nerve paralysis (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 5 | 2
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 1
Hyperreflexia (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 1
Loss of consciousness (Nervous system disorders) | 5 | 1
Neuralgia (Nervous system disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 3 | 1
Paraparesis (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Post herpetic neuralgia (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 5 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0
VIIth nerve paralysis (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 0
Hypomania (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0
Anuria (Renal and urinary disorders) | 0 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Oliguria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 4 | 4
Renal failure acute (Renal and urinary disorders) | 7 | 9
Renal impairment (Renal and urinary disorders) | 1 | 1
Ureteric obstruction (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 4
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute febrile neutrophilic dermatosis (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 3
Embolism (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 5 | 2
Hypovolaemic shock (Vascular disorders) | 3 | 0
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 9 | 1
Shock haemorrhagic (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PAN+BTZ (N=381) | PBO+BTZ (N=377)
Anaemia (Blood and lymphatic system disorders) | 154 | 125
Leukopenia (Blood and lymphatic system disorders) | 61 | 31
Lymphopenia (Blood and lymphatic system disorders) | 52 | 35
Neutropenia (Blood and lymphatic system disorders) | 112 | 40
Thrombocytopenia (Blood and lymphatic system disorders) | 238 | 150
Conjunctivitis (Eye disorders) | 28 | 31
Abdominal distension (Gastrointestinal disorders) | 30 | 25
Abdominal pain (Gastrointestinal disorders) | 50 | 38
Abdominal pain upper (Gastrointestinal disorders) | 43 | 36
Constipation (Gastrointestinal disorders) | 101 | 122
Diarrhoea (Gastrointestinal disorders) | 254 | 155
Dyspepsia (Gastrointestinal disorders) | 47 | 43
Nausea (Gastrointestinal disorders) | 137 | 78
Vomiting (Gastrointestinal disorders) | 91 | 47
Asthenia (General disorders) | 77 | 51
Fatigue (General disorders) | 155 | 109
Oedema peripheral (General disorders) | 108 | 72
Pyrexia (General disorders) | 90 | 48
Bronchitis (Infections and infestations) | 20 | 25
Herpes zoster (Infections and infestations) | 15 | 36
Nasopharyngitis (Infections and infestations) | 49 | 46
Respiratory tract infection (Infections and infestations) | 17 | 20
Upper respiratory tract infection (Infections and infestations) | 65 | 53
Urinary tract infection (Infections and infestations) | 23 | 15
Alanine aminotransferase increased (Investigations) | 22 | 19
Blood creatinine increased (Investigations) | 37 | 21
Blood urea increased (Investigations) | 20 | 10
Platelet count decreased (Investigations) | 43 | 17
Weight decreased (Investigations) | 44 | 17
Decreased appetite (Metabolism and nutrition disorders) | 106 | 46
Hyperglycaemia (Metabolism and nutrition disorders) | 30 | 25
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 | 8
Hypocalcaemia (Metabolism and nutrition disorders) | 35 | 32
Hypokalaemia (Metabolism and nutrition disorders) | 100 | 52
Hyponatraemia (Metabolism and nutrition disorders) | 48 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 42 | 32
Arthralgia (Musculoskeletal and connective tissue disorders) | 25 | 26
Back pain (Musculoskeletal and connective tissue disorders) | 45 | 46
Bone pain (Musculoskeletal and connective tissue disorders) | 21 | 31
Muscle spasms (Musculoskeletal and connective tissue disorders) | 23 | 21
Muscular weakness (Musculoskeletal and connective tissue disorders) | 24 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 24
Pain in extremity (Musculoskeletal and connective tissue disorders) | 40 | 54
Dizziness (Nervous system disorders) | 67 | 61
Dysgeusia (Nervous system disorders) | 36 | 26
Headache (Nervous system disorders) | 51 | 40
Hypoaesthesia (Nervous system disorders) | 28 | 34
Neuralgia (Nervous system disorders) | 38 | 44
Neuropathy peripheral (Nervous system disorders) | 117 | 133
Paraesthesia (Nervous system disorders) | 24 | 27
Peripheral sensory neuropathy (Nervous system disorders) | 42 | 46
Polyneuropathy (Nervous system disorders) | 28 | 28
Insomnia (Psychiatric disorders) | 73 | 61
Cough (Respiratory, thoracic and mediastinal disorders) | 81 | 70
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 53 | 40
Rash (Skin and subcutaneous tissue disorders) | 33 | 23
Hypertension (Vascular disorders) | 27 | 23
Hypotension (Vascular disorders) | 49 | 34
Orthostatic hypotension (Vascular disorders) | 22 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial